CLINICAL TRIAL: NCT02726100
Title: Systematic Medical Assessment, Referral and Treatment for Diabetes Care in China Using Lay Family Health Promoters
Brief Title: SMARTHealth Diabetes in China Using Lay Family Health Promoters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute for Global Health, China (Other)
Collaborators: Global Alliance for Chronic Diseases (GACD) (Other); National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Puhong Zhang, Associate Director, The George Institute for Global Health, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: APP1094712
Record Dates: First submitted 2016-03-22; First posted 2016-04-01 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension; Dyslipidemias
Keywords: Telemedicine; Diabetes Mellitus, Type 2; Decision Support Systems, Clinical; Family Health Promoter; Primary Health Care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Dyslipidemias

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participants in intervention communities will receive the SMARTHealth Diabetes intervention that connects community health service centers and family health providers for diabetes management. Medical staff and FHPs in the intervention communities will be provided with an initial training session on the installation and use of the platform.
  Interventions: Behavioral: SMARTHealth Diabetes
- Control arm (No Intervention): Control group doesn't use SMARTHealth Diabetes.The "usual-care" in our study will be conducted in a standard way which is defined in the Guidance of National Essential Public Health Service. All the relevant doctors in control group will be trained and required to record the activities defined in the guidance.

INTERVENTIONS:
Behavioral: SMARTHealth Diabetes — SMARTHealth Diabetes is an interactive mobile health platform to promote improved self-management for people with T2DM.
  Arms: Intervention arm

SUMMARY:
It's a community-based parallel-arm cluster Randomized Controlled Trial (RCT). An interactive mobile health management system will be developed to support lay family health promoters and healthcare staff to improve clinical outcomes for family members with Type 2 Diabetes Mellitus (T2DM). 2,000 participants from 80 sites will be chosen from urban (40 communities) and rural (40 villages) settings in Shijiazhuang City, Hebei Province.

DETAILED DESCRIPTION:
Study design and Settings:

Cluster randomised controlled trial involving 80 sites (40 communities in urban Shijiazhuang and 40 villages in rural Shijiazhuang) and 2,000 people with T2DM.

Hypothesis:

An interactive mobile health management system can support lay family health promoters (FHP) and healthcare staff to improve clinical outcomes for family members with T2DM

Intervention:

SMARTHealth Diabetes is an interactive mobile health platform to promote improved self-management for people with T2DM. It comprises the following core features:

* Management support based on best practice clinical guidelines
* Self-management tools and resources for family members
* Password protected registration of patients and their nominated FHP to access this information
* Population of key clinical information into a desktop application used by health care providers when applicable

Community eligibility:

* 40 urban communities and 40 rural villages from geographically dispersed regions will be selected
* Each community/ village must have at least one community health station providing services to ≥1,000 adult residents
* Staff at the community health station must be willing to participate in the intervention

Statistical power:

80 clusters and a mean community cluster size of 25 participants (2,000 total) will provide 90% power to detect an absolute improvement of 10% in the primary outcome. This assumes 20% of people in the control arm will achieve ≥2 'ABC' diabetes goals ((HbA1C<7%; Blood Pressure <140/80 mmHg, LDL cholesterol <100mg/dl or 2.6mmol/L) at end of study; an intra-class correlation coefficient of 0.05, a 20% loss to follow-up, and a 2-sided significance level of 0.05. This translates to a mean reduction of 0.35% for HbA1C, 0.14 mmol/L for LDL cholesterol and 3.4mmHg for systolic BP. Primary analyses will be conducted at the patient level. Secondary analyses will be conducted at the cluster level. Sub-group analyses will be conducted at the community level (based on size and health service characteristics) and patient level (based on demographic factors (co-habitation with FHP) and clinical factors (control rate of 'ABC' risk factors at baseline).

Significance:

The Chinese government has placed prevention and treatment of diabetes as one of 11 National Basic Public Health Services. Despite great promise for mobile health (mHealth) interventions to improve access to effective healthcare, there remains uncertainty about how this can be successfully achieved. These uncertainties pose substantial dilemmas for health system planners. The findings are likely to inform policy on a scalable strategy to overcome sub-optimal access to effective health care in China.

ELIGIBILITY:
Inclusion Criteria:

* Established T2DM
* HbA1C >= 7%
* Nominated family member with mobile internet access who agrees to be a family health promoter (FHP)
* Able to provide informed consent

Exclusion Criteria:

Psychologically or physically unable to participate the trials.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2073 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-10-19 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
The proportion of patients achieving at least two "ABC" goals | 24 months
  The proportion of patients achieving at least two "ABC" goals defined as any two of the following: HbA1c <7.0%, blood pressure (BP) <140/80mmHg and LDL cholesterol <100mg/dl or 2.6mmol/L) at 24 months

SECONDARY OUTCOMES:
The proportion of patients achieving the "A" goal | 24 months
  The proportion of patients achieving HbA1c <7.0% at 24 months
The proportion of patients achieving the "B" goal | 24 months
  The proportion of patients achieving blood pressure (BP) <140/80mmHg at 24 months
The proportion of patients achieving the "C" goal | 24 months
  The proportion of patients achieving LDL cholesterol <100mg/dl or 2.6mmol/L at 24 months
The proportion of patients achieving FPG<7.0 mmol/L | 24 months
  The proportion of patients achieving FPG<7.0 mmol/L at 24 months
Mean change in HbA1c level | 24 months
  Mean change in HbA1c level from baseline to 24 months
Mean changes in systolic and diastolic blood pressure levels | 24 months
  Mean changes in systolic and diastolic blood pressure levels from baseline to 24 months
Mean change in LDL cholesterol level | 24 months
  Mean change in LDL cholesterol level from baseline to 24 months
Mean change in FPG level | 24 months
  Mean change in FPG level from baseline to 24 months
Mean change in the Summary of Diabetes Self-Care Activities (SDSCA) from baseline to 24 month | 24 months
  The Summary of Diabetes Self-Care Activities is a scale to measure patients' self-management. The minimum value of each scale item is 0 and the maximum value is 7. Higher scores mean a better outcome.

OTHER OUTCOMES:
Mean change in body mass index (BMI) | 24 months
  Mean change in body mass index (BMI) from baseline to 24 months
Mean change in waist circumstance (WC) | 24 months
  Mean change in waist circumstance (WC) from baseline to 24 months
Mean change in the European quality of life 5 dimensions 3 levels scale (EQ-5D-3L) index value | 24 months
  Mean change in the European quality of life 5 dimensions 3 levels scale (EQ-5D-3L) index value from baseline to 24 months. The minimum value of the scale is 0 and the maximum value is 1. Higher scores mean a better outcome.
Mean change in the European quality of life overall self-rated visual analogue scale (EQ-VAS) | 24 months
  Mean change in the European quality of life overall self-rated visual analogue scale (EQ-VAS) from baseline to 24 months. The minimum value of the scale is 0 and the maximum value is 100. Higher scores mean a better outcome.
Mean change in The Summary of Diabetes Self-Care Activities (SDSCA) from baseline to 24 months | 24 months
  Pending
Mean change in urine albumin creatinine ratio (ACR) | 24 months
  Mean change in urine albumin creatinine ratio (ACR) from baseline to 24 months
Mean change in estimated glomerular filtration rate (GFR) | 24 months
  Mean change in estimated glomerular filtration rate (GFR) from baseline to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Puhong Zhang, PhD, Principal Investigator — The George Institute for Global Health at Peking University Health Science Center; David Peiris, PhD, Principal Investigator — The George Institute for Global Health, University of Sydney
Locations (2):
- China (2):
  - Hebei Medical University, Shijiazhuang, Hebei
  - Center of Disease Control and Prevention, Luquan, Shijiazhuang, Hebei

IPD SHARING:
Plan to Share IPD: No
Data are only accessed by investigators.

REFERENCES:
- [Derived] Tao X, Mao L, Zhang P, Ma X, Liang Z, Sun K, Peiris D. Barriers and facilitators to primary care management of type 2 diabetes in Shijiazhuang City, China: a mixed methods study. BMC Prim Care. 2024 Mar 13;25(1):84. doi: 10.1186/s12875-024-02330-7. PMID 38481166
- [Derived] Peiris D, Sun L, Patel A, Tian M, Essue B, Jan S, Zhang P. Systematic medical assessment, referral and treatment for diabetes care in China using lay family health promoters: protocol for the SMARTDiabetes cluster randomised controlled trial. Implement Sci. 2016 Aug 17;11(1):116. doi: 10.1186/s13012-016-0481-8. PMID 27535128